CLINICAL TRIAL: NCT01358149
Title: Double Blind Controlled Trial of Cocoa-based Food in Children
Brief Title: Trial of Cocoa-based Food in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10.23.NRC
Record Dates: First submitted 2011-05-13; First posted 2011-05-23 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Motor Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): cocoa-based food 1
  Interventions: Other: cocoa-based food
- Treatment 1 (Active Comparator): cocoa-based food 2
  Interventions: Other: cocoa-based food

INTERVENTIONS:
Other: cocoa-based food — single intake of cocoa-based food
  Arms: placebo
Other: cocoa-based food — Single intake of cocoa-based food
  Arms: Treatment 1

SUMMARY:
Today, there is an important lack of knowledge on child metabolism and the effects of phytochemical-rich foods, which includes fruits and vegetables and plant-derived foods. Here, the investigators will monitor the metabolism of children using minimally invasive techniques at rest, and with physical/mental activities and assess the changes associated with the intake of cocoa-based food.

ELIGIBILITY:
Inclusion Criteria:

All subjects must comply with all the following inclusion criteria:

* Healthy and physically active, and no diabetes or metabolism related disorders in their first degree relatives (as determined by medical and activity questionnaire)
* Caucasian, with English as a first language and an adequate standard of literacy.
* BMI adjusted for age and gender which falls between the 9th and 91st as shown in the Child Growth Foundation BMI growth charts
* 8-13 years of age
* Having obtained his/her informed assent
* Having obtained his/her legal representative's informed consent
* Willing to allow their family doctor (GP) to be informed about their participation in this study

Exclusion Criteria:

Subjects representing one or more of the following criteria are excluded from participation in the study.

* Post-pubertal
* Taking any medication
* Smoker
* Undergoing medical treatment or investigations
* Body mass index > 24
* Suffer from chronic diseases (with regular intake of drugs, medical history)
* Vegetarians
* Vaccination in the last 4 months
* Any know food allergies or intolerance
* Pregnancy
* Special diet or weight loss program (e.g. Atkins diet)
* Acute illness
* Fever, cold, flu
* Participation in a cholesterol management program with functional foods like food supplement enriched in omega-3 fatty acids, dairy products enriched with phytosterols (margarines, yoghurts).

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Blood glucose concentration | Baseline will be fasting, and monitoring measures up to 7 hours after consumption
  Time Frame: the effects of one-off consumption will be measured over a 7-8 hours period. Baseline will be fasting, and monitoring measures up to 7 hours after consumption. The subjects will be on controlled diet the day prior to the visit.

SECONDARY OUTCOMES:
Metabolic monitoring | measured over a 7-8 hours period
  Time Frame: the effects of one-off consumption will be measured over a 7-8 hours period. Baseline will be fasting, and monitoring measures up to 7 hours after consumption. The subjects will be on controlled diet the day prior to the visit.
physical monitoring | two hours and four hours after concumption
  Time Frame: the effects of one-off consumption will be measured two hours and four hours after consumption with 45 min physical activity sessions.
mental monitoring | 3.3 hours after intake
  Time Frame: the effects of one-off consumption will be measured around 3.3 hours after intake. Baseline will be at fasting before intake.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Atkin, Prof. Dr., Principal Investigator — Hull University
Locations (1):
- Hull York Medical School, Hull, United Kingdom